CLINICAL TRIAL: NCT07241650
Title: Postoperative Pain and Quality of Life in Root Canal Treatment: Prospective Study
Brief Title: Evaluation of the Effects of Different Irrigation Solutions and Activation Methods on Postoperative Pain and Quality of Life in Root Canal Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Selen Yusufoğlu, assoc prof, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-13-19
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Irreversible Acute Pulpitis; Root Canal Treatment
Keywords: root canal irrigation; irrigation activation systems; EDDY; laser
MeSH Terms: interventions — Therapeutic Irrigation; Sodium Hypochlorite; Lasers, Semiconductor; Etidronic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the bioistatician performing the data analysis will be blinded to group allocation. the cinician performing th treatments will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sodium Hypochlorite and Conventional Syringe (Experimental): Each canal will be irrigated with 5 ml of saline for 30 seconds, followed by 10 ml of 2.5% sodium hypochlorite delivered manually using a conventional syringe, without any additional activation technique.
  Interventions: Procedure: Irrigation with Sodium Hypochlorite and Conventional Syringe
- Sodium Hypochlorite and EDDY (Experimental): Each canal will be irrigated with 5 ml of saline for 30 seconds, followed by 10 ml of 2.5% sodium hypochlorite activated for 30 seconds using the EDDY sonic device.
  Interventions: Procedure: Irrigation with Sodium Hypochlorite and EDDY
- Sodium Hypochlorite and Diode Laser (Experimental): Each canal will be irrigated with 5 ml of saline for 30 seconds, followed by 10 ml of 2.5% sodium hypochlorite activated for 30 seconds using a diode laser.
  Interventions: Procedure: Procedure: Irrigation with Sodium Hypochlorite and Diode Laser
- Etidronic Acid (HEDP) and Conventional Syringe (Experimental): Each canal will be irrigated with 5 ml of saline for 30 seconds, followed by 10 ml of HEDP (Dual Rinse) solution delivered manually using a conventional syringe, without any additional activation technique
  Interventions: Procedure: Procedure: Irrigation with Etidronic Acid and Conventional Syringe
- Etidronic Acid (HEDP) and EDDY (Experimental): Each canal will be irrigated with 5 ml of saline for 30 seconds, followed by 10 ml of HEDP (Dual Rinse) solution activated for 30 seconds using the EDDY sonic device.
  Interventions: Procedure: Procedure: Irrigation with Etidronic Acid and EDDY
- Etidronic Acid (HEDP) and Diode Laser (Experimental): Each canal will be irrigated with 5 ml of saline for 30 seconds, followed by 10 ml of HEDP (Dual Rinse) solution activated for 30 seconds using a diode laser.
  Interventions: Procedure: Irrigation with Etidronic Acid and Diode Laser

INTERVENTIONS:
Procedure: Irrigation with Sodium Hypochlorite and Conventional Syringe — Procedure: Irrigation with Sodium Hypochlorite and Conventional SyringeIn the final irrigation protocol, 5 ml of saline solution will be applied for 30 seconds, followed by 10 ml of 2.5% sodium hypochlorite delivered manually using a standard needle without any additional activation technique. Participants will be instructed to record their postoperative pain using the Visual Analogue Scale (VAS) before treatment and at 6, 12, 24, 36, 48, and 72 hours, as well as 1 week after treatment and at 6, 12, 24, 36, 48, and 72 hours, as well as 1 week after treatment. Additionally, they will complete the Oral Health Impact Profile questionnaire (OHIP-14) to assess the impact on quality of life.
  Other Names: NaOCl activated with Conventional Syringe
  Arms: Sodium Hypochlorite and Conventional Syringe
Procedure: Irrigation with Sodium Hypochlorite and EDDY — Procedure: Irrigation with Sodium Hypochlorite and EDDYSodium hypochloride with EDDY Activation In the final irrigation protocol, 5 ml of saline solution will be applied for 30 seconds, followed by 10 ml of 2.5% sodium hypochlorite, which will be activated with EDDY for 10 seconds. Each canal will receive three cycles of 10-second EDDY activation. Participants will be instructed to record their postoperative pain using the Visual Analogue Scale (VAS) before treatment and at 6, 12, 24, 36, 48, and 72 hours, as well as 1 week after treatment and at 6, 12, 24, 36, 48, and 72 hours, as well as 1 week after treatment. Additionally, they will complete the Oral Health Impact Profile questionnaire (OHIP-14) to assess the impact on quality of life.
  Other Names: NaOCl activated with EDDY
  Arms: Sodium Hypochlorite and EDDY
Procedure: Procedure: Irrigation with Sodium Hypochlorite and Diode Laser — Procedure: Irrigation with Sodium Hypochlorite and Diode LaserSodium Hypochloride with Diode Laser Activation In the final irrigation protocol, 5 ml of saline solution will be applied for 30 seconds, followed by 10 ml of 2.5% sodium hypochlorite, which will be activated with a diode laser for 10 seconds. Each canal will receive three cycles of 10-second laser activation. Participants will be instructed to record their postoperative pain using the Visual Analogue Scale (VAS) before treatment and at 6, 12, 24, 36, 48, and 72 hours, as well as 1 week after treatment and at 6, 12, 24, 36, 48, and 72 hours, as well as 1 week after treatment. Additionally, they will complete the Oral Health Impact Profile questionnaire (OHIP-14) to assess the impact on quality of life.
  Other Names: NaOCl activated with Diode Laser
  Arms: Sodium Hypochlorite and Diode Laser
Procedure: Procedure: Irrigation with Etidronic Acid and Conventional Syringe — Procedure: Irrigation with Etidronic Acid and Conventional SyringeEtidronic Acid with Conventional Syringe In the final irrigation protocol, 5 ml of saline solution will be applied for 30 seconds, followed by 10 ml of 2.5% sodium hypochlorite mixed with HEDP, delivered manually using a standard needle without additional activation. Participants will be instructed to record their postoperative pain using the Visual Analogue Scale (VAS) before treatment and at 6, 12, 24, 36, 48, and 72 hours, as well as 1 week after treatment and at 6, 12, 24, 36, 48, and 72 hours, as well as 1 week after treatment. Additionally, they will complete the Oral Health Impact Profile questionnaire (OHIP-14) to assess the impact on quality of life.
  Other Names: HEDP with Conventional Syringe
  Arms: Etidronic Acid (HEDP) and Conventional Syringe
Procedure: Procedure: Irrigation with Etidronic Acid and EDDY — Etidronic Acid with EDDY Activation In the final irrigation protocol, 5 ml of saline solution will be applied for 30 seconds, followed by 10 ml of 2.5% sodium hypochlorite mixed with HEDP, which will be activated with EDDY for 10 seconds. Each canal will receive three cycles of 10-second EDDY activation. Participants will be instructed to record their postoperative pain using the Visual Analogue Scale (VAS) before treatment and at 6, 12, 24, 36, 48, and 72 hours, as well as 1 week after treatment. Additionally, they will complete the Oral Health Impact Profile questionnaire (OHIP-14) to assess the impact on quality of life.
  Other Names: HEDP with EDDY
  Arms: Etidronic Acid (HEDP) and EDDY
Procedure: Irrigation with Etidronic Acid and Diode Laser — Etidronic Acid with Diode Laser Activation In the final irrigation protocol, 5 ml of saline solution will be applied for 30 seconds, followed by 10 ml of 2.5% sodium hypochlorite mixed with HEDP, which will be activated with a diode laser for 10 seconds. Each canal will receive three cycles of 10-second laser activation. Participants will be instructed to record their postoperative pain using the Visual Analogue Scale (VAS) before treatment and at 6, 12, 24, 36, 48, and 72 hours, as well as 1 week after treatment. Additionally, they will complete the Oral Health Impact Profile questionnaire (OHIP-14) to assess the impact on quality of life.
  Other Names: HEDP with diode laser
  Arms: Etidronic Acid (HEDP) and Diode Laser

SUMMARY:
Brief Summary: This prospective randomized controlled clinical trial aims to evaluate the effects of different irrigation solutions (NaOCl, HEDP) and activation methods (conventional syringe irrigation, EDDY, diode laser) on postoperative pain and oral health-related quality of life in single-visit root canal treatment of asymptomatic mandibular molars.

DETAILED DESCRIPTION:
The primary aim of this prospective randomized controlled clinical trial is to evaluate the effects of two different irrigation solutions (2.5% NaOCl and HEDP) and three different activation methods (conventional syringe, EDDY, diode laser) on postoperative pain and oral health-related quality of life in single-visit root canal treatment of asymptomatic mandibular molars, aiming to overcome the limitations of conventional irrigation. Additionally, the study will compare patients' oral health-related quality of life before treatment and one week after treatment. While no significant difference in postoperative pain is expected, an improvement in quality of life is anticipated.Eligible participants will be adult patients requiring endodontic treatment of asymptomatic mandibular molars. After meeting inclusion criteria and providing informed consent, participants will be randomly assigned to six different groups. Randomization will be performed using a computer-generated random number sequence and the codes will be kept in sealed opaque envelopes to prevent bias between groups.The irrigation protocols and activation methods to be applied in the study are as follows:Irrigation Solutions: 2.5% NaOCl and HEDP (HEDP; Dual Rinse, Medcem GmbH, Weinfelden,Switzerland)Activation Techniques: Conventional syringe, EDDY (Micron, Tokyo, Japonya), diode laser Dentsply Sirona Sirolaser Advance; Sirona Dental Systems, Bensheim, Germany)Anesthesia: Regional mandibular block using Articaine-containing MaxicainAll procedures will be performed under rubber dam isolation. Root canal working length will be determined using a #10 K-type file and apex locator, and canals will be shaped using a nickel-titanium rotary system. Each canal will be irrigated according to the assigned protocol, and root canals will be obturated using gutta-percha and an epoxy resin-based sealer with a single-cone technique. Postoperative radiographs will be taken to confirm obturation, and definitive restorations will be completed with composite resin materials.Postoperative pain will be assessed using the Visual Analog Scale (VAS) at 6, 12, 24, 36, 48, 72 hours, and one week after treatment. Quality of life will be measured using the OHIP-14 questionnaire before treatment and one week postoperatively.The study sample size is 90 participants, with 15 volunteers per group. All treatments will be performed by a single operator, and the materials and devices used in the study are standard products routinely used in clinical practice. The expected benefit of the study is to determine the effects of different irrigation solutions and activation methods on postoperative pain and patient quality of life, providing insights for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Systemic Inclusion Criteria1. Volunteers must not have any systemic symptoms or be pregnant.2. According to the ASA classification, individuals with: • ASA I (Healthy (without acute and/or chronic diseases)• ASA II (with mild systemic diseases) (asymptomatic congenital heart disease, well-controlled dysrhythmias, non-exacerbated asthma, well-controlled epilepsy, non-insulin-dependent diabetes mellitus, oncological conditions in remission) will be included in our study.3. Must be between 18 and 65 years of age.4. Must not have used analgesic anti-inflammatory drugs in the last two weeks or cortisone in the last 6 months.5. Volunteers must be able to contact us again 6, 12, 24, 48, or 72 hours after completing their treatment and must be mentally fit enough to express pain scores and answer the questionnaire.6. Volunteers must not have bruxism.Local inclusion criteria 1. Mandibular molars must be present.2. Teeth must be asymptomatic preoperatively.There must be no palpation, percussion, or radiographic findings.3. Rubber dams must be attached to the teeth to be treated.4. The teeth must be in its normal position within the mouth.5. The volunteer must be able to open their mouth sufficiently.

Exclusion Criteria:

* 1. Volunteers who have used analgesics, anti-inflammatory drugs, antibiotics, etc. that could alter pain and infection control in the last 12 hours.2. Subjects with a history of sensitivity or adverse reactions to any medication or material used in this study3. Teeth with calcified canals or severe periodontal disease4. Subjects with missing opposing or adjacent teeth5. Pregnant or breastfeeding female subjects6. Teeth requiring additional anesthesia methods (e.g., intrapulpal, intraligamentary, second block anesthesia, or additional local anesthetic agent) will be excluded from the study if anesthesia is insufficient.7. Teeth with apical lesions will not be included in the study.8. Teeth with root resorption will not be included in the study.9. Teeth requiring restorations such as endocrowns, onlays, overlays, or full crowns due to excessive material loss after root canal treatment will not be included in the study.Teeth with structural loss sufficient to require post-core application will be excluded.10. Teeth with untreated periodontitis and teeth or sites that have undergone surgical treatment within the last 6 months will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
VAS scala | 6., 12.,24.,36.,48.,72 hours and 1 week
  VAS (Visual Analog Scale): As its name suggests, the visual analog scale (VAS) uses an analog format, representing a continuous range of values. The most common way to measure pain on a VAS is with a 10 cm (100 mm) horizontal line. The volunteer is asked to place a mark on this line, which is then measured and recorded in millimeters or centimeters.According to the VAS scale, they will mark the pain they feel before treatment and after 6, 12, 24, 36, 48, 72 hours and 1 week (VAS) on the form.
OHIP test | 7 days
  (OHIP14) Scale will be asked to be filled before treatment and one week after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt Universty, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peters OA, Schonenberger K, Laib A. Effects of four Ni-Ti preparation techniques on root canal geometry assessed by micro computed tomography. Int Endod J. 2001 Apr;34(3):221-30. doi: 10.1046/j.1365-2591.2001.00373.x. PMID 12193268
- [Background] Scrimshaw SV, Maher C. Responsiveness of visual analogue and McGill pain scale measures. J Manipulative Physiol Ther. 2001 Oct;24(8):501-4. doi: 10.1067/mmt.2001.118208. PMID 11677548
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- [Background] Layton G, Wu WI, Selvaganapathy PR, Friedman S, Kishen A. Fluid Dynamics and Biofilm Removal Generated by Syringe-delivered and 2 Ultrasonic-assisted Irrigation Methods: A Novel Experimental Approach. J Endod. 2015 Jun;41(6):884-9. doi: 10.1016/j.joen.2015.01.027. Epub 2015 Mar 6. PMID 25749254
- [Background] Tungsawat P, Arunrukthavorn P, Phuntusuntorn P, Opatragoon S, Sirirangsee P, Inklub S. Comparison of the Effect of Three Irrigation Techniques and Root Canal Preparation Size on Sodium Hypochlorite Penetration into Root Canal Dentinal Tubules. Int J Dent. 2021 Mar 31;2021:6612588. doi: 10.1155/2021/6612588. eCollection 2021. PMID 33859692
- [Background] Rosier RN, O'Keefe RJ. Autocrine regulation of articular cartilage. Instr Course Lect. 1998;47:469-75. No abstract available. PMID 9571448
- [Background] Heerema NA, Sather HN, Sensel MG, Lee MK, Hutchinson RJ, Nachman JB, Reaman GH, Lange BJ, Steinherz PG, Bostrom BC, Gaynon PS, Uckun FM. Abnormalities of chromosome bands 13q12 to 13q14 in childhood acute lymphoblastic leukemia. J Clin Oncol. 2000 Nov 15;18(22):3837-44. doi: 10.1200/JCO.2000.18.22.3837. PMID 11078497
- [Background] Perdigao P. Definitions and treatment regimens for recurrent tuberculosis. Int J Tuberc Lung Dis. 2000 Apr;4(4):384-5. No abstract available. PMID 10777091
- [Background] Udrea E, Dancau N. [Idiopathic pulmonary hemosiderosis (2 clinical cases)]. Rev Ig Bacteriol Virusol Parazitol Epidemiol Pneumoftiziol Pneumoftiziol. 1977 Jul-Sep;26(3):185-8. Romanian. PMID 201012